CLINICAL TRIAL: NCT05823116
Title: A Randomized Clinical Trial of Continuous vs. Intermittent Infusion Vancomycin: Effects on Measured GFR and Kidney Injury Biomarkers
Brief Title: Continuous vs. Intermittent Infusion Vancomycin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aaron Cook (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Aaron Cook, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83412; R21AI176298 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Vancomycin
Keywords: Infusion; Adverse Effect; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin continuous infusion (Active Comparator): Continuous infusion of Vancomycin
  Interventions: Drug: Vancomycin Continuous Infusion
- Vancomycin intermittent infusion (Active Comparator): Intermittent infusion of vancomycin
  Interventions: Drug: Vancomycin Intermittent Infusion

INTERVENTIONS:
Drug: Vancomycin Continuous Infusion — A precision drug dosing platform will be used to determine the empiric dosing regimen and the dosing parameter targeted will be an area-under-the-curve (AUC) of 500 mg⸱hr/L (range 400-600 mg⸱hr/L). The total daily dose is infused over a period of 24 hours.
  Other Names: Vancocin
  Arms: Vancomycin continuous infusion
Drug: Vancomycin Intermittent Infusion — A precision drug dosing platform will be used to determine the empiric dosing regimen and the dosing parameter targeted will be an area-under-the-curve (AUC) of 500 mg⸱hr/L (range 400-600 mg⸱hr/L). The dose is infused at rates of 1 gram per hour in every 8, -12, or -24 hour intervals.
  Other Names: Vancocin
  Arms: Vancomycin intermittent infusion

SUMMARY:
Hospitalized adult participants prescribed vancomycin by their treating physician will be randomized to receive vancomycin via continuous or intermittent infusion and measures of kidney function and injury will be collected.

DETAILED DESCRIPTION:
All study participants regardless of participation status will have been prescribed vancomycin by a treating physician and received a dose per institutional standard of care. Participants will be randomized 1:1 in permuted blocks of 2, 4, or 6 to receive subsequent doses via continuous or intermittent infusion. Participants randomized to intermittent infusion will receive doses per standard of care at infusion rates of 1 gram per hour in every 8,-12, or -24 hour intervals, while participants randomized to continuous infusion will receive a total daily dose infused over a period of 24 hours.

Vancomycin concentration will not exceed 5mg/ml and will be infused via central (preferred) or peripheral administration. In order to ensure consistent dosing between study arms, a precision dosing platform will be used by the PI and team to determine total daily doses to best target an AUC of 500 mg x hr/L (range 400-600 mg x hr/L). A single vancomycin concentration will be obtained the following day with Bayesian-guided area-under-the-curve (AUC) monitoring (with dosing adjusted if needed) to ensure vancomycin exposure remains similar between infusion strategies. Both the initiation and discontinuation of vancomycin, as well as any additional therapeutic drug monitoring, will remain at the discretion of the primary clinical team.

Glomerular filtration rate (GFR) will be measured on the day of enrollment and day 3 by the administration of 5 ml iohexol (300 mgI/ml) with iohexol plasma concentrations obtained 1 and 4 hours following administration of iohexol. This change in measured GFR between the infusion strategies is the primary outcome of the study. Plasma and urinary markers of kidney function and injury will be obtained the day of enrollment (Day 0) and subsequent days (Days 2-3). If the participant remains on vancomycin 120 hours following enrollment, measured glomerular filtration rate (mGFR) and biomarkers will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Hospitalized at University of Kentucky on a medical service (internal medicine or medical intensive care)
* Prescribed ≥ 2 doses of vancomycin per treating physician
* Be able to provide written, informed consent, or have a legally authorized representative (LAR) responsible for their care able to provide written, informed consent.

Exclusion Criteria:

* Chronic kidney disease (documented or prior to admission estimated GFR (eGFR) <60 ml/min/1.73m2 using non-race-based creatinine GFR equation)
* End stage kidney disease
* Stage 1 or higher AKI per Kidney Disease: Improving Global Outcomes (KDIGO) classification (serum creatinine increase ≥ 0.3 mg/dl or 1.5-1.9 times baseline; urine output < 0.5 ml/kg/hr for 6-12 hours)
* Greater than 2 doses of vancomycin within the last 72 hours
* Allergy to iohexol
* Uroepithelial tumors
* Pregnancy
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Change in measured glomerular filtration rate (GFR) | Baseline (Day 0) and Day 3
  measured via the administration of a small dose of iohexol followed by the collection of blood samples
Change in urinary Kidney Injury Molecule 1 (KIM-1) | Baseline (Day 0) and Day 3
  Measured by urine ELISA test as the change score

SECONDARY OUTCOMES:
Plasma cystatin C over time | Baseline up to 5 days
  Measured by urine ELISA test at baseline, 48-, and 72-hours following the first dose of vancomycin.
  Additional measure at 120 hours if the patient is prescribed vancomycin for 120 hours or more.
Urine Clusterin over time | Baseline up to 5 days
  Measured by urine ELISA test at baseline, 48-, and 72-hours following the first dose of vancomycin. Additional measure at 120 hours if the patient is prescribed vancomycin for 120 hours or more.
Urine Osteopontin over time | Baseline up to 5 days
  Measured by urine ELISA test at baseline, 48-, and 72-hours following the first dose of vancomycin. Additional measure at 120 hours if the patient is prescribed vancomycin for 120 hours or more.
Urine Kidney Injury Molecule-1 (KIM-1) over time | Baseline up to 5 days
  Measured by urine ELISA test test at baseline, 48-, and 72-hours following the first dose of vancomycin. Additional measure at 120 hours if the patient is prescribed vancomycin for 120 hours or more.
Change in Urine Kidney Injury Molecule-1 (KIM-1) | Baseline (Day 0) and Day 5
  Measured as the change score, only in the only in subset of patients prescribed 5 or more days of vancomycin
Vancomycin Area-Under-the-Curve (AUC) target attainment | Day 1
  Defined as range 400-600 mg*hr/L. AUC assessed using one concentration Bayesian estimates.
Acute Kidney Injury (AKI) over time | Daily up to 10 days
  Using serum creatinine and urine output components of Kidney Disease: Improving Global Outcome (KIDGO) classification
Phlebitis over time | Daily up to 7 days
  Monitored per standard of care, using phlebitis scores of 0 (no clinical symptoms) to 4. Documented scores above 0 will be classified as phlebitis.
Infiltration over time | Daily up to 7 days
  Monitored per standard of care, using infiltration scores of 0 (no clinical symptoms) to 4. Documented scores above 0 will be classified as infiltration.
Acute Kidney Disease | Until hospital discharge, up to 17 days
  measured per Acute Disease Quality Initiative (ADQI) criteria in a subset of participants where AKI does not resolve by 7 days
Number of Participants with Major Adverse Kidney Events | Until hospital discharge, up to 17 days
  Composite of death, requirement for kidney replacement therapy, or reduction of 25% from baseline estimated glomerular filtration rate.
Change in measured glomerular filtration rate (GFR) | Baseline (Day 0) and Day 5
  measured via the administration of a small dose of iohexol followed by the collection of blood samples, only in the subset of patients receiving vancomycin for 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Cook, PharmD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT05823116/ICF_000.pdf